CLINICAL TRIAL: NCT05811988
Title: Cost Assessment of Videolaryngoscopy Compared to Direct Laryncoscopy in a Large Academic Center
Status: Completed | Type: Observational
Sponsor: Adam Thaler (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Sponsor
Other Study IDs: VL vs DL cost
Record Dates: First submitted 2022-10-18; First posted 2023-04-13 (Actual); Last update posted 2023-04-13 (Actual); Status verified 2023-04

CONDITIONS: Economic Problems

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Direct Laryngoscopy
- Video Laryngoscopy

SUMMARY:
Cost, both direct and indirect, assessment of videolaryngoscopy, specifically the McGrath, compared to direct laryncoscopy in a large academic center.

ELIGIBILITY:
Data were obtained on all endotracheal intubations where the Anesthesiology service was assigned to staff a surgical case requiring tracheal intubation during general anesthesia. Data were also obtained for tracheal intubations outside the operating room (ICUs, Trauma, patient wards) when Anesthesiology personnel were requested which did not include the Emergency Department

Electronic patients' medical records spanning a two-year period (July 1, 2019 to June 30, 2021)

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Adults
Sampling Method: Probability Sample
Enrollment: 66987 (Actual)
Dates: Start 2022-03-31 (Actual); Primary Completion 2022-06-15 (Actual); Study Completion 2022-06-15 (Actual)

PRIMARY OUTCOMES:
Cost comparison | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Thomas Jefferson University, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
Plan to publish